CLINICAL TRIAL: NCT04071938
Title: Shared Responsibility Between General Practitioners and Highly Specialized Hospitals in Complex Chronic Conditions: the Case of Spinal Cord Injury in a Nationwide Intervention Study
Brief Title: Shared Responsibility Between General Practitioners and Highly Specialized Hospitals in Spinal Cord Injury
Acronym: SCICO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Schweizer Paraplegiker Forschung (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: SCICO
Record Dates: First submitted 2019-08-26; First posted 2019-08-28 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): Physicians: 10 GPs from 10 practices who treat patient with Spinal cord injury (SCI) and 10 SCI specialists.
  Patients: 270 people with SCI within 25 minutes vehicle driving distance to the GP practices will be in the intervention group
  Interventions: Other: Teaching to GPs; Other: Site visits to GP practices
- Control group (No Intervention): Physicians: 20 GPs who treat patient with SCI will not receive any intervention. They will be completing the questionnaire (DOC) and assessed for satisfaction with collaboration with the SCI specialist.
  Patients: 210 people with spinal cord injury outside the catchment area of the intervention group will be receiving usual care (no intervention)

INTERVENTIONS:
Other: Teaching to GPs — Educational modules on bladder, bowel and skin-care, and pain management will be provided to participating GPs by Spinal Cord Injury specialists
  Arms: Intervention group
Other: Site visits to GP practices — Visits by specialized nurses to the participating GPs at their practices to support the establishment of specialized care on-site
  Arms: Intervention group

SUMMARY:
It is an interventional study that aims to assess a new primary care model of collaboration between specialized centers and primary care physicians in Switzerland, in order to reduce morbidity and improve patients' and providers' experience with delivery of follow-up care in individuals with chronic spinal cord injury as compared to current best practice.

DETAILED DESCRIPTION:
This model will lead to awareness, recognition and interactive communication between GPs and specialists and guidelines on the shared-role relationship.

The study interventions are educational modules on bladder, bowel, skin-care, and pain management which will be provided to participating GPs by Spinal Cord Injury specialists. In addition visits by specialized nurses to the participating GPs at their practices to support the establishment of specialized care on-site.

ELIGIBILITY:
Inclusion Criteria:

Physicians

* GPs practicing in medium to large group practice
* The practice is wheelchair accessible and remote to SCI specialized centers
* Proficiency certificate in ultrasonography

Patients:

* Diagnosed with traumatic or non-traumatic, sensory or motor complete or incomplete, chronic SCI
* 18 years or older
* Permanently reside in Switzerland
* Reside farther than 25 minutes driving distance from a specialized SCI center
* Understand German, English, Italian
* Informed consent
* Additionally in treatment group: Patients with chronic SCI Living in the region of a participating GP irrespective if they visit the participating primary care practice.
* Additionally in control group: individuals with SCI who live outside the catchment areas

Exclusion Criteria:

Patients:

- Acute SCI or during first rehabilitation phase - Congenital conditions leading to paraplegia or tetraplegia, including spina bifida - Neurodegenerative disorders such as multiple sclerosis and amyotrophic lateral sclerosis - Guillain-Barré syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 273 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Average difference in total score of Doctor's Opinions on Collaboration (DOC) | Change from baseline to 12 and 24 months post intervention
  DOC is a validated questionnaire covering organization, communication, professional expertise, image and knowing each other. It will be completed by GPs and SCI specialists. The DOC will be converted to an interval score and scaled from 0 to 100 with minimum and maximum score (0=completely agree, 100=completely disagree)
Average difference in total score of Modified Spinal Cord Injury Secondary Conditions Scale (SCI-SCS) score | Change from baseline to 12 and 24 months post intervention
  Modified Spinal Cord Secondary Conditions Scale (SCI-SCS) targets secondary conditions associated with SCI composite endpoint, excluding diabetes mellitus and joint and muscle pain. Modified (SCI-SCS) includes 14 health conditions and chronic pain. Self reporting through questionnaires on pressure sores, urinary tract infections, spasticity, postural hypotension, bowel, and bladder problems, etc...). The rating scale uses a 4-point ordinal scale ranging from 0 (not experienced/insignificant problem never limiting activity) to 3 (significant/chronic problem).

SECONDARY OUTCOMES:
Physicians' satisfaction | Change in overall satisfaction scores from baseline to 12 and 24 months post intervention
  Questionnaire distributed to physicians in intervention and control group to measure the difference in the satisfaction with the collaboration between the health care providers.
Average difference in the number of inpatient hospitalization | Change from baseline to 12 months and 24 months post intervention
  Number of hospitalizations people with SCI had in 12 months period
Average difference in number of patients visits to a specialist or a SCI center | Change from baseline to 12 and 24 months post intervention
  Number of visits to SCI specialist of SCI center people with SCI had in 12 months period
Average difference in subscore on pressure sores | Change from baseline to 12 and 24 months post intervention
  from Modified Spinal Cord Injury Secondary Conditions Scale (SCI-SCS)Subscore on pressure sores with a 4-point rating on severity, ranging from 0 (not experienced/insignificant problem never limiting activity) to 3 (significant/chronic problem)
Average difference in subscore on UTIs | Change from baseline to 12 and 24 months post intervention
  from Modified Spinal Cord Injury Secondary Conditions Scale (SCI-SCS)Subscore on urinary tract infections (UTIs) with a 4-point rating on severity, ranging from 0 (not experienced/insignificant problem never limiting activity) to 3 (significant/chronic problem)

CONTACTS AND LOCATIONS:
Overall Officials: Armin Gemperli, PhD, Principal Investigator — Schweizer Paraplegiker Forschung
Locations (1):
- Schweizer Paraplegiker Forschung, Nottwil, Canton of Lucerne, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tomaschek R, Touhami D, Essig S, Gemperli A. Shared responsibility between general practitioners and highly specialized physicians in chronic spinal cord injury: Study protocol for a nationwide pragmatic nonrandomized interventional study. Contemp Clin Trials Commun. 2021 Nov 17;24:100873. doi: 10.1016/j.conctc.2021.100873. eCollection 2021 Dec. PMID 34869940